CLINICAL TRIAL: NCT02659124
Title: Comparison of AmnioFix Laser and Standard of Care in Patients Seeking Laser Facial Treatment
Brief Title: Comparison of AmnioFix Laser and Standard of Care Treatment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The current protocol did not satisfy IRB requirements
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AmnioFix Laser Study
Record Dates: First submitted 2016-01-11; First posted 2016-01-20 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Rhytides
Keywords: facial laser; fraction ablative resurfacing; total ablative resurfacing; EpiFix; rhytides; wrinkles; AmnioFix
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Standard of Care plus AmnioFix (Other): All patients will receive the standard of care alone on half of their face, and AmnioFix in addition to the standard of care on the other half of their face.
  Interventions: Device: AmnioFix plus Standard of Care; Procedure: Standard of Care

INTERVENTIONS:
Device: AmnioFix plus Standard of Care — Patients will receive the standard of care alone on half of their face, and AmnioFix in addition to the standard of care on the other half of their face. The standard of care after ablative resurfacing is conservative wound care which may include flexible wound care dressings and/or emollients.
Procedure: Standard of Care — Patients will receive the standard of care dressing only, on their face. The standard of care after ablative resurfacing is conservative wound care which may include flexible wound care dressings and/or emollients.

SUMMARY:
This is a comparison trial with novel application of AmnioFix and a control arm. Patients electively being treated with facial lasers will be assigned to receive AmnioFix in addition to the normal standard of care placed on half of their face after laser procedure, and normal post laser standard of care alone on the other half of their face. The investigators will investigate the end points of healing, recovery time, re-epitheliaziation, and other cosmetic factors. The study is designed to compare AmnioFix to the current standard of laser care.

DETAILED DESCRIPTION:
AmnioFix is a dehydrated Human Amnion/ Chorion Membrane (dHACM) allograft and is composed of multiple layers including a single layer of epithelial cells, a basement membrane and an avascular connective tissue matrix. Amniotic membrane is a unique material and its composition contains collagen types I, III, IV, V, and VII. Amniotic membrane is composed of structural extracellular matrix (ECM), that also contains specialized proteins fibronectin, laminins, proteoglycans and glycosaminoglycans. In addition, amniotic membrane contains essential, active, healing growth factors such as epidermal growth factor (EGF), transforming growth factor beta (TGF-b), fibroblast growth factor (FGF), and platelet derived growth factor (PDGF).

The study is designed to compare AmnioFix to the current standard of laser care.

* Patients coming in for fraction or total ablative resurfacing with any methods will be studied
* patients will be assessed prior to any treatment by clinician
* additionally patients will participate in a clinician constructed survey
* patients will be assessed on a rating scale of 1-4 based on erythema, edema/induration, oozing/drainage, and epithelialization
* preoperative photos will be taken of patients
* laser resurfacing will proceed under clinician guidance, and under clinician selected settings
* repeat photographs
* patients will be randomized as to which side of the face receives AmnioFix treatment, and which side receives standard of care
* epifix will be applied appropriatly
* repeat photographs and repeat assessment on 1-4 scale
* patients will follow up at day 1, 4, 7, 14, and 28 +/-3 days to repeat scoring and photography

ELIGIBILITY:
Inclusion Criteria:

* adult patients ages 18-100 seeking laser facial treatment

Exclusion Criteria:

* patients with treatment areas with active or latent infection
* patient with a disorder that would create an unacceptable risk of post-operative complications

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2017-04 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Time of reepithelialization | 28 days after treatment
  Subjects' healing and recovery is the primary outcome measure. Reepithelialization will be assessed at each follow up visit, considering the following: erythema, edema/induration, and oozing/drainage.

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF Dermatology, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No